CLINICAL TRIAL: NCT06213207
Title: Saving Lives of Newborn (SaLiN): A Cluster Randomized Controlled Trial Applying Helping Baby Breathe to Manage Birth Asphyxia in Sarlahi District of Madhesh Province, Nepal
Brief Title: Cluster Randomized Controlled Trial Applying Helping Baby Breathe in Nepal
Acronym: SaLiN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrated Development Foundation Nepal (Other)
Collaborators: Women and Children Welfare Society Nepal (Unknown)
Responsible Party: Principal Investigator, Khem Pokhrel, Dr. Khem Pokhrel, Principal Investigator, SaLiN Project, Integrated Development Foundation Nepal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NP593-2023; 2023-0091 (Other Grant/Funding Number: Laerdal Foundation)
Record Dates: First submitted 2023-12-29; First posted 2024-01-19 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Newborn Morbidity; Newborn Asphyxia; Delivery Preterm
Keywords: Skilled birth attendant; Management of newborn asphyxia; Neonatalie; Cluster Randomized Controlled Trial; Nepal
MeSH Terms: conditions — Asphyxia Neonatorum; Premature Birth

STUDY DESIGN:
Intervention Model Description: The intervention is targeted to provide simulator based training to newborn care service providers. The training is comprised of essential newborn care practices and the providers will be followed up and provided mentoring and coaching for the period of six months.
Who Masked: Outcomes Assessor
Masking Description: As this is a cluster randomized controlled trial, masking is not possible. The intervention participants from intervention cluster receive intervention and control will be receiving usual services. The outcomes assessor will not be known about the name of health facilities. This is done using coding of the health facilities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newborn care service providers with simulation-based training and newborns (Experimental): Newborn care providers will be the subject for receiving intervention. The will receive 5 days training on managing essential newborn care and birth asphyxia using neonatalie. The service providers will be provided monthly mentoring and coaching. The newborn who receive the services
  Interventions: Other: Simulator based training to manage asphyxia and essential newborn care using neonatalie
- Controlled health facilities with newborn care service providers with no training and newborns (No Intervention): The newborn care providers from control health facilities will not receive any additional training. They provide usual services.

INTERVENTIONS:
Other: Simulator based training to manage asphyxia and essential newborn care using neonatalie — The intervention, HBB training package will be used which was applied to train the hospitals staff in Nepal (Chaulagain et al., 2021) and Laerdal Global Health (Laerdal Global Health, 2021) to enhance the competencies on the resuscitation to newborn using NeoNatalie. Health workers will receive 5 days simulation training by expert pediatrician and pediatric nurse who have prior working experience in Neonatal Intensive Care Unit (NICU) or Special Neonatal Care Unit. After the training, mentoring and coaching will be provided experienced newborn coach/trainer on a monthly basis for six months.
  Arms: Newborn care service providers with simulation-based training and newborns

SUMMARY:
The cluster randomized controlled trial will be conducted in the selected health facilities/birthing centers of Sarlahi district in Nepal. Further from the selected health facilities. The investigators will assess the newborn in terms of their health outcomes. Characteristics related to the performance of skilled birth attendants will be measured prior to the intervention. After six months of the intervention, endline assessment will be conducted. The intervention unit are the health facilities which provide the services as birthing centers. The effectiveness of the intervention will be examined using generalized estimating equation against baseline vs. endline on skills performance of the health workers and newborn health outcomes. The study will be implied in the similar settings to improve the skill performance and newborn health outcomes in order to reduce neonatal mortality.

DETAILED DESCRIPTION:
In Nepal, health facilities need to be strengthened and the staff should be tailored training at health facilities who are designated as birthing center. Although, the health facility readiness survey has shown that health facilities had availability of bag and mask (neonatal) neonatal resuscitation equipment in delivery room (Kc et al., 2020). However, health workers were found to have lack of adequate knowledge on basic emergency and neonatal care (BEmONC) signal function including poor knowledge and skill on newborn resuscitation. resulting in poor child health outcomes during facility-births and had poor knowledge and skill on newborn resuscitation (Lama et al., 2020). Newborn resuscitation simulation training was effective in improving clinical performance of health service providers and perinatal outcomes (Vadla, Moshiro, et al., 2022). NeoNatalie™ is a low-cost, highly portable, and realistic manikin that helps health workers learn and practice standard newborn care and resuscitation measures to better handle birth asphyxia(Laerdal helping save lives, 2022). Use of NeoNatalie, a newborn simulator for neonatal resuscitation training has improved performance of midwives and their motivation(Vadla, Mdoe, et al., 2022). There has been intervention that provided training on helping baby breathe (HBB) in large hospitals in Nepal. However, the use of simulator and training to the midwives at birthing center has not been evaluated for the effectiveness of simulator in increasing their performance and newborn health outcomes. Therefore, this study aimed to improve the performance of skilled-birth attendant in providing resuscitation to the newborn with birth asphyxia by applying simulator-based training.

ELIGIBILITY:
Inclusion Criteria

Health service providers those are directly involved in providing newborn care services

Have received Community-based Integrated Management of Neonatal and Childhood Illness (CB-IMNCI) training Have worked in the study facilities at least one year

Exclusion Criteria:

Health workers, Those lack experience at least six months of working in birthing centers Those who does not qualify as skilled birth attendant (non-SBA) Those who received training already

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-18 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Skill performance of the newborn care provider | six months
  The skill performance of the newborn care providers covering all nine components of essential newborn care. Their skills related to resuscitation procedures will be measured using skill inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Adhikari, MD, Study Chair — Kanti Children's Hospital, Kathmandu
Locations (1):
- Development and Research Service International Nepal, Lalitpur, Nepal

IPD SHARING:
Plan to Share IPD: No